CLINICAL TRIAL: NCT05471349
Title: Message Testing in Older Adult Smokers (MCAS-2)
Brief Title: Message Testing in Older Adult Smokers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Centiment LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-0624; 1K23AG067929-01A1 (NIH); 2022-0624 (Other: UW Madison); A534253 (Other: UW Madison); SMPH/MEDICINE/GEN INT MD (Other: UW Madison)
Record Dates: First submitted 2022-07-20; First posted 2022-07-22 (Actual); Results first posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Smoking; Smoking Cessation
MeSH Terms: conditions — Smoking; Smoking Cessation | interventions — Videotape Recording

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hope message (Active Comparator): Participants will view a hope-based video message and flyer.
  Interventions: Behavioral: Flyer and video
- Fear message (Active Comparator): Participants will view a fear-based video message and flyer.
  Interventions: Behavioral: Flyer and video
- Control message (Placebo Comparator): Participants will view a water advertisement video and flyer.
  Interventions: Behavioral: Flyer and video

INTERVENTIONS:
Behavioral: Flyer and video — Participants will view a flyer and video

SUMMARY:
This study is examining different messages to motivate older smokers to quit smoking. Participants will be current smokers, between the ages of 50-80 years old, who do not have a history of cognitive impairment or dementia. Participants can expect to take part in a one-time 30 minute online survey.

ELIGIBILITY:
Inclusion Criteria:

* Current smoker (smoking at least some days per week)
* Ability to read and write English
* Between the ages of 50 and 80 years old

Exclusion Criteria:

* History of Mild Cognitive Impairment or dementia

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 820 (Actual)
Dates: Start 2022-07-12 (Actual); Primary Completion 2022-07-18 (Actual); Study Completion 2022-07-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adrienne Johnson, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hope Message | Fear Message | Control Message
Started | 280 | 274 | 266
Completed | 280 | 272 | 264
Not Completed | 0 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hope Message | Fear Message | Control Message | Total
Number analyzed (Participants) | 280 | 274 | 266 | 820
Age, Customized [Mean (Standard Deviation); unit: years] | 60.90 (7.456) | 61.13 (7.606) | 61.19 (7.180) | 61.07 (7.411)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  cisgender man | 133 | 129 | 134 | 396
  cisgender woman | 135 | 137 | 122 | 394
  Non-binary | 3 | 1 | 3 | 7
  transgender man | 0 | 1 | 0 | 1
  transgender woman | 0 | 0 | 1 | 1
  other | 6 | 4 | 4 | 14
  refuse to answer | 3 | 2 | 2 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 6 | 17 | 31
  Not Hispanic or Latino | 270 | 267 | 249 | 786
  Unknown or Not Reported | 2 | 1 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 7 | 7 | 9 | 23
  Asian | 7 | 4 | 8 | 19
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 69 | 68 | 54 | 191
  White | 182 | 182 | 182 | 546
  More than one race | 7 | 9 | 8 | 24
  Unknown or Not Reported | 8 | 3 | 5 | 16
Region of Enrollment [Number; unit: participants]
  United States | 280 | 274 | 266 | 820

OUTCOME MEASURES:

1. Primary Outcome: Emotional Response
Description: Measure participants' emotional response to the messages using a 1-9 scaled measurement of 14 different emotions (9 indicating more emotional response). Emotionality will be presented together summarizing the mean presentation of these emotions by the different groups.
Time Frame: Through study completion, approximately 30 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hope Message | Fear Message | Control Message
Number analyzed (Participants) | 280 | 272 | 264
score on a scale
  Felt sad | 2.73 (2.231) | 2.97 (2.363) | 1.26 (1.066)
  Felt angry | 2.17 (2.026) | 2.04 (1.862) | 1.26 (1.1221)
  Felt afraid | 2.74 (2.302) | 2.98 (2.443) | 1.31 (1.100)
  Felt guilty | 3.14 (2.500) | 3.30 (2.604) | 1.32 (1.224)
  Felt disgusted | 2.33 (2.221) | 2.37 (2.210) | 1.36 (1.328)
  Felt worried | 3.18 (2.525) | 3.60 (2.584) | 1.39 (1.222)
  Felt ashamed | 2.83 (2.418) | 2.66 (2.317) | 1.32 (1.215)
  Felt confused | 1.94 (1.755) | 1.76 (1.679) | 1.47 (1.397)
  Felt amused | 2.15 (1.987) | 2.10 (1.977) | 3.91 (2.548)
  Felt hopeful | 4.53 (2.628) | 4.37 (2.606) | 4.41 (2.610)
  Felt motivated | 4.42 (2.561) | 4.26 (2.614) | 4.34 (2.803)
  Felt understood | 5.09 (2.719) | 5.18 (2.753) | 4.82 (2.809)
  Felt happy | 3.20 (2.425) | 2.68 (2.331) | 5.13 (2.573)
  Felt surprised | 3.28 (2.547) | 3.10 (2.563) | 3.24 (2.546)

2. Primary Outcome: Motivation to Quit
Description: Measure participants' motivation to quit after viewing the flyer and video, using a 1 item scaled measurement of motivation to quit (1-7 scale, 7 indicating higher motivation).
Time Frame: Through study completion, approximately 30 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Hope Message | Fear Message | Control Message
Number analyzed (Participants) | 280 | 272 | 264
score on a scale | 4.20 (1.917) | 3.93 (1.999) | 3.93 (2.003)

ADVERSE EVENTS:
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed due to the minimal risk, single interaction, brief duration (~15mins), online survey extent of the study procedures.
Arm/Group | Hope Message | Fear Message | Control Message
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2023-12-11): https://cdn.clinicaltrials.gov/large-docs/49/NCT05471349/Prot_000.pdf